CLINICAL TRIAL: NCT04827407
Title: Lipopolysaccharide Adsorption At Septic Shock with Efferon LPS Extracorporeal Blood Adsorbers
Brief Title: Lipopolysaccharide Adsorption At Septic Shock
Acronym: LASSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Collaborators: Ligand Research, LLC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-lps-2021-01
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Septic Shock
Keywords: septic shock; extracorporeal therapy; LPS adsorption; abdominal sepsis
MeSH Terms: conditions — Shock, Septic; Intraabdominal Infections

STUDY DESIGN:
Intervention Model Description: A multicentre randomised clinical trial evaluating the efficacy and safety of the Efferon LPS device in extracorporeal hemoperfusion in patients with abdominal sepsis complicated with septic shock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic therapy + Efferon LPS (Experimental): Basic therapy is the institution's routine practice for treating patients with septic shock against a background of abdominal sepsis plus extracorporeal hemoperfusion therapy (Efferon LPS)
  Interventions: Device: Efferon LPS hemoperfusion
- Baseline therapy (No Intervention): Basic therapy is the institution's routine practice for treating patients with septic shock against a background of abdominal sepsis.

INTERVENTIONS:
Device: Efferon LPS hemoperfusion — Hemoperfusion using continuous extracorporeal LPS adsorption with Efferon LPS therapeutic device during a period of 24h immediately following admission to the intensive care unit
  Other Names: extracorporeal blood adsorption
  Arms: Basic therapy + Efferon LPS

SUMMARY:
Sepsis is a global healthcare burden sepsis, it reaches 20-30 million cases annually (WHO data). Numerous studies have shown that extracorporeal hemoperfusion therapies that eliminate endotoxin and\or excess of cytokines improve treatment outcomes in patients with septic shock. The main purpose of the study is to obtain new data on the efficacy and safety of the Efferon LPS device in extracorporeal therapy in patients with abdominal sepsis complicated by septic shock.

DETAILED DESCRIPTION:
Sepsis is a global healthcare burden sepsis, it reaches 20-30 million cases annually (WHO data). A two-stage trial by Rudnov et al. using one-day data from 62 centres in 29 subjects of the Russian Federation showed that one third of the patients admitted to the ICU were patients with infection, one fifth of them developed septic shock, the proportion of hospital sepsis was 46.6%, and fatal outcome occurred in 30.4% of patients with infection. Despite apparent advances in intensive care, the prognosis of patients with endotoxaemia and septic shock remains poor.

Extracorporeal removal of toxic substances from the bloodstream by adsorbing them onto a porous material may provide clear clinical benefits. Extracorporeal blood adsorption method can be a good complement or substitute for the classical methods of haemofiltration and haemodialysis if the diffusion or convection of toxic substances through the membrane is not efficient enough. Since the method was first proposed by Muirhead and Reid in 1948, it has developed considerably.

Endotoxin (lipopolysaccharide), one of the most potent mediators of sepsis, is found in high concentrations in about 50% of patients with septic shock. The use of extracorporeal sorption techniques that eliminate endotoxin has been shown in numerous trials to improve outcomes in patients with septic shock.

Efferon LPS (Efferon JSC, Moscow, Russia) is a single-use therapeutic device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by selective adsorption of lipopolysaccharides (bacterial endotoxins) and non-selective removal of cytokines by internal porous structure. It is a cylindrical polycarbonate casing filled with spherical granules of LPS-selective polymeric adsorbent mesoporous beads and isotonic sodium chloride solution. The device is registered in Russia as a medical device RZN 2019/8886.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Established diagnosis of Gram-negative septic shock according to SEPSIS-3 criteria
* The immediate post-operative period (no more than 24 hours after surgery)
* Hypotension requiring vasopressor support: the need for at least one of the vasopressors listed below at the dose listed below for at least 2 hours continuously and not more than 12 hours.

  * Norepinephrine> 0.05 µg/kg/min
  * Dopamine> 10 µg/kg/min
  * Phenylephrine> 0.4 µg/kg/min
  * Adrenaline > 0.05 µg/kg/min
  * Vasopressin> 0.03 units/min Vasopressin (any dose) in combination with another vasopressor listed above
* The patient must have received intravenous infusion therapy of at least 30 ml/kg administered within 24 hours of inclusion.
* The patient's condition allows therapy with the Efferon LPS device for at least 4 hours.

Exclusion Criteria:

Lack of adequate antimicrobial chemotherapy

* Identifying the criteria for non-inclusion;
* A patient may voluntarily withdraw from a trial at any time after giving informed consent and before the trial is completed. The investigator may also withdraw a participant from the trial at any time at his or her discretion and for any of the following reasons:
* Reasons for a participant's withdrawal from the trial will be recorded and may include, amongst others, the following
* Withdrawal of consent to participate in the trial by the participant.
* The development of an adverse event, including a serious one; individual intolerance to the investigational product, hypersensitivity to the components of the product due to which further participation in the trial is not possible.
* Continued participation in the trial is not, in the researcher's opinion, in the participant's health interests.
* The presence of deviations from the plan which, in the opinion of the Sponsor and Investigator, require the withdrawal of the participant from the trial.
* A positive pregnancy test result at any time during the test.
* When any participant withdraws from a trial, the reason for the withdrawal should be documented.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Effect of the Efferon LPS hemoperfusion in extracorporeal therapy in patients with abdominal sepsis complicated by septic shock | 1-14 days
  The time (number of days) from randomisation to the earliest time that the 'resolution of septic shock' event is achieved. Event criteria: 1) end of vasopressor support (persistence of effect - for 4 hours) and 2) investigator/trained staff rating the trial as 'resolved' when assessed from baseline to day 14 or hospital discharge (if discharge occurs earlier than day 14).

SECONDARY OUTCOMES:
Effect of the Efferon LPS hemoperfusion on systemic haemodynamic parameters after the start of use in patients with abdominal sepsis complicated by septic shock | 1-72 hours
  Sats every 6 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours. The time (number of days) from randomisation to the end of vasopressor support within 72 x hours or hospital discharge (if earlier than 72 hours). Maximum dose of vasopressors within 24 hours and 72 hours of the start of hemoperfusion.
Effect of the Efferon LPS hemoperfusion on pulmonary oxygen metabolism function in patients with abdominal sepsis complicated by septic shock | 1-72 hours
  Value of oxygenation index (Pa02 / Fi02 (Pa) every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours
Effect of the Efferon LPS hemoperfusion on the length of stay in the ICU of patients with abdominal sepsis complicated by septic shock | 1-14 days
  The time (number of days) from randomisation to transfer from the ORIT within 14 days or hospital discharge or transfer from the ORIT (if occurring earlier than day 14).

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Rey, MD, PhD, Principal Investigator — N. V. Sklifosovsky Moscow Research Institute of Emergency, Moscow, Russia; Vladimir Kulabukhov, MD, PhD, Principal Investigator — N. V. Sklifosovsky Moscow Research Institute of Emergency, Moscow, Russia
Locations (4):
- Russia (4):
  - V.P. Demikhov City Clinical Hospital No. 68, Moscow
  - N.I. Pirogov City Clinical Hospital No. 1, Moscow
  - N.V. Sklifosovsky Moscow Research Institute of Emergency, Moscow
  - S.S. Yudin City Clinical Hospital, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rey S, Kulabukhov VM, Popov A, Nikitina O, Berdnikov G, Magomedov M, Kim T, Masolitin S, Ignatenko O, Krotenko N, Marysheva A, Chaus N, Ohinko L, Mendibaev M, Chumachenko A, Pisarev V. HEMOPERFUSION USING THE LPS-SELECTIVE MESOPOROUS POLYMERIC ADSORBENT IN SEPTIC SHOCK: A MULTICENTER RANDOMIZED CLINICAL TRIAL. Shock. 2023 Jun 1;59(6):846-854. doi: 10.1097/SHK.0000000000002121. Epub 2023 Apr 6. PMID 37018802
- [Background] Ushakova N.D., Tikhonova S.N., Rozenko D.A. Hemosorption by a Column Adsorber Based on Hyper-Cross-Linked Styrene-Divinylbenzene Copolymer with Immobilized Lipopolysaccharide-Selective Ligand in Combined Intensive Care of Lung Cancer-Related Postoperative Acute Lung Injury (Case Report). General Reanimatology. 2020;16(4):14-20. https://doi.org/10.15360/1813-9779-2020-4-14-20
- [Background] Magomedov M.A., Kim T.G., Masolitin S.V., Yaralian A.V., Kalinin E.Yu., Pisarev V.M. Use of Sorbent Based on Hypercrosslinked Styrene-Divinylbenzene Copolymer With Immobilized LPS-Selective Ligand In Hemoperfusion For Treatment of Patients With Septic Shock. General Reanimatology. 2020;16(6):31-53. https://doi.org/10.15360/1813-9779-2020-6-31-53
- See also: https://doi.org/10.15360/1813-9779-2020-4-14-20 — https://doi.org/10.15360/1813-9779-2020-4-14-20
- See also: https://doi.org/10.15360/1813-9779-2020-6-31-53 — https://doi.org/10.15360/1813-9779-2020-6-31-53
- See also: https://doi.org/10.21320/1818-474X-2023-4-60-71 — https://doi.org/10.21320/1818-474X-2023-4-60-71